CLINICAL TRIAL: NCT07323953
Title: Prospective Clinical Trial Evaluating AmblyoFix for the Treatment of Unilateral Amblyopia in Children
Brief Title: Evaluation of AmblyoFix for the Treatment of Unilateral Amblyopia in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eyesight Electronics (Industry)
Collaborators: Al Watany Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFX-PCT-EG-2025
Record Dates: First submitted 2025-12-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Amblyopia
Keywords: Amblyopia Treatment
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AmblyoFix (Experimental): Participants assigned to this arm will undergo binocular vision therapy using the AmblyoFix software on a laptop, in combination with red-blue anaglyph glasses. Prior to therapy initiation, a calibration process will be completed and validated by the study team to ensure device screen specifications meet protocol requirements. Treatment consists of interactive, gamified visual tasks designed to stimulate the amblyopic eye under binocular viewing conditions.
  Interventions: Behavioral: AmblyoFix binocular digital therapy

INTERVENTIONS:
Behavioral: AmblyoFix binocular digital therapy — AmblyoFix is a binocular vision therapy delivered through specialized software on a laptop computer in combination with red-blue anaglyph glasses. The program uses interactive, gamified visual tasks designed to stimulate the amblyopic eye while maintaining binocular viewing conditions. Each participant undergoes a standardized calibration process to ensure screen specifications are validated before starting therapy.

SUMMARY:
This is a prospective, single-arm, non-inferiority clinical trial designed to evaluate the efficacy, safety, and adherence of AmblyoFix binocular digital therapy for the treatment of unilateral amblyopia in children aged 7 to 12 years. Outcomes will be compared against a retrospective cohort of patients of the same age range previously treated with standard occlusion (patching) at the same clinic.

A total of 33 participants will be enrolled, allowing for up to 15% attrition to ensure at least 28 evaluable completers at Week 24. Eligible participants must have unilateral amblyopia with amblyopic-eye best-corrected visual acuity (BCVA) between 0.3 and 1.3 logMAR and an interocular difference of at least 0.2 logMAR, with stable refractive correction for at least 16 weeks prior to enrollment.

The primary outcome is the change in amblyopic-eye BCVA (logMAR) from baseline to Week 24, assessed under standardized Snellen or ETDRS protocol by certified, masked outcome assessors. Secondary outcomes include adherence (captured via in-software usage logs), safety (BCVA worsening ≥2 lines and ocular adverse events), and patient-reported outcomes (acceptability, usability, satisfaction). An interim analysis will be conducted at Week 6 and at Week 12 to review early efficacy and safety, with the option to recommend early termination if robust evidence of non-inferiority is demonstrated.

In addition to the primary study population of unilateral amblyopia, an exploratory subgroup of 3 or more participants with bilateral amblyopia may be enrolled for observational evaluation. Treatment will initially target the eye with worse BCVA as selected in the AmblyoFix software. Upon sufficient improvement, as determined by the Principal Investigator, treatment may be switched to the other eye within the software settings. Data from the bilateral exploratory cohort will be analyzed descriptively and reported separately. These data will not contribute to the primary non-inferiority analysis.

Participants and caregivers cannot be blinded due to the nature of the intervention; however, outcome assessors and statisticians will remain masked to study objectives and comparator data to minimize bias. Follow-up assessments will occur at baseline, Week 6, Week 12, and Week 24, with no additional amblyopia treatment permitted during the study unless clinically required.

This trial is designed to rigorously determine whether AmblyoFix is a safe, effective, and non-inferior alternative to patching, with the potential to improve adherence, usability, and acceptability in real-world amblyopia therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-12 years.
* Unilateral amblyopia secondary to anisometropia and/or mild strabismus.
* BCVA in amblyopic eye between 20/40-20/400 (0.3-1.3 logMAR); fellow eye ≥20/32 (≤0.2 logMAR).
* Interocular difference ≥2 lines (≥0.2 logMAR).
* Stable refractive correction for ≥16 weeks or <0.1 logMAR change across two visits ≥8 weeks apart.
* Cycloplegic refraction within 7 months meeting anisometropia criteria (e.g., hyperopia ≥+2.50 D).
* Access to a suitable home environment (laptop and internet).
* Parent/guardian consent and child assent (7+ year olds).

Exclusion Criteria:

* Atropine use within 2 weeks before starting treatment
* Prior amblyopia treatment beyond refractive adaptation.
* Myopia >-6.00 D SE, previous ocular surgery, or other ocular pathology.
* Severe cognitive/developmental delay impeding compliance.
* History of light-induced seizures.
* Inability/unwillingness to comply with digital monitoring.
* Any condition compromising safety or trial integrity.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Change in BCVA in the amblyopic eye from baseline to Week 24 | From enrollment to the end of treatment at 24 Weeks
  The primary outcome of this trial is the change in best-corrected visual acuity (BCVA) in the amblyopic eye from baseline to week 24, measured in logMAR units using the Snellen or ETDRS protocol. This approach was selected for its clinical validity, reproducibility, and alignment with international standards in amblyopia trials. Visual acuity will be assessed monocularly under best optical correction, with the fellow eye occluded during testing. Certified, masked outcome assessors will conduct all measurements in standardized conditions to minimize bias, with testing procedures (including lighting, calibration, and display specifications) harmonized.

SECONDARY OUTCOMES:
Adherence to AmblyoFix | From enrollment to the end of treatment at 24 Weeks
  Adherence will be objectively measured through the AmblyoFix software's built-in time-tracking functions, which automatically record session frequency and duration. Adherence will be calculated as the total minutes of active use per week compared with the prescribed target duration. Mean weekly adherence will be derived over the 24-week treatment period.
  Unit of Measure: Total minutes of active use per week (minutes/week)
Safety of Amblyofix | From enrollment to the end of treatment at 24 Weeks
  Safety will be evaluated by recording all adverse events (AEs) and serious adverse events (SAEs) throughout the 24-week intervention period. Particular attention will be paid to ocular health, including reports of visual discomfort, diplopia, or any unexpected effects potentially related to digital therapy or occlusion. All safety data will be reviewed and summarized by the study investigators at each follow-up visit and at study completion. Unit of Measure: Number of participants with adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Watany Research and Development Center, Watany Eye Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No